CLINICAL TRIAL: NCT05565157
Title: Flapless Zygomatic Implants Robot-assisted Placement
Acronym: ROSA-ZYGOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0076
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Zygomatic Implant; Robotic
Keywords: zygomatic implant; robotic; flapless; mini-invasive; ROSA; immediate loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Zygomatic implants — A robotic assisted new strategy for positioning zygomatic implants will be performed and its efficacy and accuracy will be assess

SUMMARY:
Zygomatic implants are indicated for the rehabilitation of the severely atrophic maxilla. Similar to standard implant placement, gaining an optimal position of the zygomatic implants is essential for a predictable prosthetic-driven treatment outcome.

However, there is no effective mechanism to physically control the drilling trajectory for the zygomatic implants. Therefore, deviation between the actual and planned implant position is inevitable.

This approach is technically difficult, and is performed by an experienced surgeon.

The development of a surgical technique that is both safer and less invasive is currently possible thanks to robotics. In this project, a robotic assisted new strategy for positioning zygomatic implants will be performed and its efficacy and accuracy will be assess.

Path planning will be carried out on a pre-operative scanner. The ROSA robot (Zimmer®) will guide the several drillings steps. Placement of the zygomatic implant will be performed manually.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Maxillary edentulism with severe bone resorption
* Patients suffering from maxillary edentulism post maxillary defect (carcinologic or traumatic) and free flap reconstruction
* Patients suffering from post-maxillectomy buccosinusal communication.
* Age ≥ 18 years old
* Having signed the informed consent

Exclusion Criteria:

* Patients suffering from chronic sinusitis
* Patients refusing ROSA robot-guided surgery (unsigned informed consent).
* Pregnant and nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Variation rate between theoretical intraoperative position and post-operative zygomatic implants position | one day
  The accuracy of zygomatic implants positioning will be evaluated by comparing the theoretical intraoperative position and the actual post-operative position by image fusion.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No